CLINICAL TRIAL: NCT04315181
Title: Prescription Medications: Pharmacodynamics and Interaction Effects
Brief Title: Prescription Medication Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sharon Walsh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Walsh, Director, Center on Drug and Alcohol Research, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 46591; R01DA016718 (NIH)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use; Sedative Use
Keywords: opioid; sedative; opiate
MeSH Terms: interventions — Analgesics, Opioid; Hypnotics and Sedatives

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a randomized, double-blind, double-dummy, placebo- controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Placebo / Placebo (Placebo Comparator): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Placebo / Oxycodone 20mg (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Placebo / Oxycodone 40mg (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Gabapentin 600mg / Placebo (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Gabapentin 1200mg / Placebo (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Gabapentin 600mg / Oxycodone 20mg (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Gabapentin 1200mg / Oxycodone 20mg (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Gabapentin 600mg / Oxycodone 40mg (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives
- Gabapentin 1200mg / Oxycodone 40mg (Experimental): Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Interventions: Drug: Opioid Agonist; Drug: Sedatives

INTERVENTIONS:
Drug: Opioid Agonist — Abuse liability evaluation.
Drug: Sedatives — Abuse liability evaluation.

SUMMARY:
This study will examine the effects of doses of opioid/placebo and doses of sedative/placebo, alone and in combination. The primary outcomes are related to pharmacodynamic measures (subjective ratings of drug liking and other abuse-related effects; physiological outcomes) to determine the interaction effects of these compounds.

DETAILED DESCRIPTION:
Gabapentin and oxycodone are commonly used in combination for the treatment of chronic pain. Gabapentin is now widely misused/abused with studies indicating that gabapentin abuse is especially common among individuals with opioid misuse. The nature of gabapentin's abuse-related effects have been described in case reports and online as sedative-like and opioid-like, with descriptive reports including sedation, euphoria, talkativeness and increased energy. Despite their widespread co-administration both for licit and illicit purposes, no controlled psychopharmacological studies to our knowledge have directly examined the effects of oxycodone (or another opioid agonist) and gabapentin in combination. This study's objective is to characterize the subjective effect profile of gabapentin, examine the interaction between gabapentin and oxycodone, and assess the acute analgesic response to gabapentin and oxycodone, alone and in combination, across a range of doses for each drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, ages 18-55
* Current non-medical use of opioids and sedatives

Exclusion Criteria:

* Physical dependence on opioids, alcohol, or benzodiazepines/sedatives/hypnotics
* Seeking treatment for drug use
* Significant medical problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Walsh, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Center on Drug and Alcohol Research, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover study with 9 conditions tested in random order in each completing subject.
Groups:
- Prescription Medication Interactions: Within subject study. Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Opioid Agonist: Active opioid agonist or placebo, administered orally
  Sedatives: Active sedative or placebo, administered orally
Period: Overall Study
Arm/Group | Prescription Medication Interactions
Started | 11
Placebo/Placebo | 10
Placebo / Oxycodone 20mg | 10
Placebo / Oxycodone 40mg | 10
Gabapentin 600mg / Placebo | 10
Gabapentin 1200mg / Placebo | 10
Gabapentin 600mg / Oxycodone 20mg | 10
Gabapentin 1200mg / Oxycodone 20mg | 10
Gabapentin 600mg / Oxycodone 40mg | 10
Gabapentin 1200mg / Oxycodone 40mg | 10
Completed | 10
Not Completed | 1
Not completed — Non-responsive to drug conditions. | 1

BASELINE CHARACTERISTICS:
Population: One participant did not complete the study. They were non-responsive to the drug conditions and was discharged.
Groups:
- Completing Participants: Subjects who completed the full study (i.e., completed all dose conditions) Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Opioid Agonist: Active opioid agonist or placebo, administered orally
  Sedatives: Active sedative or placebo, administered orally
Arm/Group | Completing Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.80 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Subject-Rated Outcome: Visual Analog Scale (VAS) Drug Liking
Description: Participants rated their subjective drug liking on a standardized VAS scale (0 to 100). Raw data transformed to peak scores. Higher scores indicate greater drug effects.
Time Frame: This outcome was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session).
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo / Placebo | Placebo / Oxycodone 20mg | Placebo / Oxycodone 40mg | Gabapentin 600mg / Placebo | Gabapentin 1200mg / Placebo | Gabapentin 600mg / Oxycodone 20mg | Gabapentin 1200mg / Oxycodone 20mg | Gabapentin 600mg / Oxycodone 40mg | Gabapentin 1200mg / Oxycodone 40mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Score on a scale | 7.40 (2.39) | 39.00 (7.19) | 40.80 (9.14) | 24.50 (8.54) | 15.00 (8.70) | 40.70 (9.10) | 34.50 (8.26) | 56.50 (6.85) | 44.90 (8.29)
Statistical Analysis 1: Comparison: Placebo / Placebo vs Placebo / Oxycodone 20mg vs Placebo / Oxycodone 40mg vs Gabapentin 600mg / Placebo vs Gabapentin 1200mg / Placebo vs Gabapentin 600mg / Oxycodone 20mg vs Gabapentin 1200mg / Oxycodone 20mg vs Gabapentin 600mg / Oxycodone 40mg vs Gabapentin 1200mg / Oxycodone 40mg; Peak scores were calculated for individual participants within each dose condition and analyzed in a one-factor model (drug condition) with a compound symmetry covariance structure; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Statistical significance is 2-sided and accepted at a P value of ≤ 0.05; F=6.89, df=8, 72

2. Secondary Outcome: Change in Subject-Rated Outcome: Visual Analog Scale (VAS) Drug Effect
Description: Participants rated their subjective drug effect on a standardized VAS scale (0 to 100). Raw data transformed to peak scores. Higher scores indicate greater drug effects.
Time Frame: as for outcome 1
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Placebo / Oxycodone 40mg: Participants will receive non-therapeutic experimental doses of gabapentin (600 and 1200 mg, p.o.), alone and in combination with oxycodone (20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
  Sedatives: Active sedative or placebo, administered orally
Arm/Group | Placebo / Placebo | Placebo / Oxycodone 20mg | Placebo / Oxycodone 40mg | Gabapentin 600mg / Placebo | Gabapentin 1200mg / Placebo | Gabapentin 600mg / Oxycodone 20mg | Gabapentin 1200mg / Oxycodone 20mg | Gabapentin 600mg / Oxycodone 40mg | Gabapentin 1200mg / Oxycodone 40mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Score on a scale | 10.70 (2.94) | 39.30 (6.32) | 39.70 (8.05) | 25.00 (7.43) | 21.50 (9.93) | 39.10 (7.37) | 37.50 (7.73) | 52.30 (8.36) | 44.40 (8.51)
Statistical Analysis 1: Comparison: Placebo / Placebo vs Placebo / Oxycodone 20mg vs Placebo / Oxycodone 40mg vs Gabapentin 600mg / Placebo vs Gabapentin 1200mg / Placebo vs Gabapentin 600mg / Oxycodone 20mg vs Gabapentin 1200mg / Oxycodone 20mg vs Gabapentin 600mg / Oxycodone 40mg vs Gabapentin 1200mg / Oxycodone 40mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Statistical significance is 2-sided and accepted at a P value of ≤ 0.05; F=5.51, df=8, 72

3. Secondary Outcome: Change in Respiration Rate
Description: Respiration rate (number of breaths per minute). Raw data transformed to trough scores. Lower scores indicate greater impairment.
Time Frame: Respiration rate was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session).
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: Number of breaths per minute
Arm/Group | Placebo / Placebo | Placebo / Oxycodone 20mg | Placebo / Oxycodone 40mg | Gabapentin 600mg / Placebo | Gabapentin 1200mg / Placebo | Gabapentin 600mg / Oxycodone 20mg | Gabapentin 1200mg / Oxycodone 20mg | Gabapentin 600mg / Oxycodone 40mg | Gabapentin 1200mg / Oxycodone 40mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Number of breaths per minute | 12.70 (0.68) | 12.00 (0.42) | 11.50 (0.54) | 12.10 (0.41) | 12.90 (0.66) | 11.80 (0.51) | 12.10 (0.59) | 11.30 (0.47) | 11.90 (0.57)
Statistical Analysis 1: Comparison: Placebo / Placebo vs Placebo / Oxycodone 20mg vs Placebo / Oxycodone 40mg vs Gabapentin 600mg / Placebo vs Gabapentin 1200mg / Placebo vs Gabapentin 600mg / Oxycodone 20mg vs Gabapentin 1200mg / Oxycodone 20mg vs Gabapentin 600mg / Oxycodone 40mg vs Gabapentin 1200mg / Oxycodone 40mg; Trough scores were calculated for individual participants within each dose condition and analyzed in a one-factor model (drug condition) with a compound symmetry covariance structure; Test type: Superiority; p = 0.138, Mixed Models Analysis — Statistical significance is 2-sided and accepted at a P value of ≤ 0.05; F=1.61, df=8, 72

4. Secondary Outcome: Change in End-tidal Carbon Dioxide (EtCO2)
Description: EtCO2 collected via capnograph monitored throughout each session. Raw data transformed to peak scores. Higher scores indicate greater impairment.
Time Frame: EtCO2 recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session).
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: mm Hg (unit of pressure)
Arm/Group | Placebo / Placebo | Placebo / Oxycodone 20mg | Placebo / Oxycodone 40mg | Gabapentin 600mg / Placebo | Gabapentin 1200mg / Placebo | Gabapentin 600mg / Oxycodone 20mg | Gabapentin 1200mg / Oxycodone 20mg | Gabapentin 600mg / Oxycodone 40mg | Gabapentin 1200mg / Oxycodone 40mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
mm Hg (unit of pressure) | 39.60 (1.01) | 41.20 (0.87) | 42.90 (1.08) | 39.10 (0.64) | 38.40 (0.48) | 42.00 (0.75) | 41.90 (0.59) | 44.80 (0.68) | 43.90 (0.90)
Statistical Analysis 1: Comparison: Placebo / Placebo vs Placebo / Oxycodone 20mg vs Placebo / Oxycodone 40mg vs Gabapentin 600mg / Placebo vs Gabapentin 1200mg / Placebo vs Gabapentin 600mg / Oxycodone 20mg vs Gabapentin 1200mg / Oxycodone 20mg vs Gabapentin 600mg / Oxycodone 40mg vs Gabapentin 1200mg / Oxycodone 40mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Statistical significance is 2-sided and accepted at a P value of ≤ 0.05; F=8.15, df=8, 72

5. Secondary Outcome: Change in Oxygen Saturation
Description: Oxygen saturation (measured as a percentage through pulse ox) monitored throughout each session. Raw data transformed to trough scores. Lower scores indicate greater impairment.
Time Frame: Oxygen saturation recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session).
Population: Per Protocol population, defined as participants completing the 9 experimental drug conditions.
Measure: Mean (Standard Error); unit: Percentage of oxygen in blood
Arm/Group | Placebo / Placebo | Placebo / Oxycodone 20mg | Placebo / Oxycodone 40mg | Gabapentin 600mg / Placebo | Gabapentin 1200mg / Placebo | Gabapentin 600mg / Oxycodone 20mg | Gabapentin 1200mg / Oxycodone 20mg | Gabapentin 600mg / Oxycodone 40mg | Gabapentin 1200mg / Oxycodone 40mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Percentage of oxygen in blood | 96.77 (0.40) | 96.29 (0.25) | 95.72 (0.53) | 96.86 (0.58) | 96.87 (0.32) | 96.59 (0.19) | 96.29 (0.28) | 95.80 (0.45) | 95.61 (0.41)
Statistical Analysis 1: Comparison: Placebo / Placebo vs Placebo / Oxycodone 20mg vs Placebo / Oxycodone 40mg vs Gabapentin 600mg / Placebo vs Gabapentin 1200mg / Placebo vs Gabapentin 600mg / Oxycodone 20mg vs Gabapentin 1200mg / Oxycodone 20mg vs Gabapentin 600mg / Oxycodone 40mg vs Gabapentin 1200mg / Oxycodone 40mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0002, Mixed Models Analysis — Statistical significance is 2-sided and accepted at a P value of ≤ 0.05; F=4.58, df=8, 72

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks. AE monitoring begins once consent is signed and is tracked through participant disqualification or follow-up visit.
Description: Adverse event definitions are the same as the clinicaltrials.gov definitions.
Groups:
- Pre-Intervention / Days Off: Prior to any drug administration or on participant days off when AE is not related to drug conditions.
- Qualification: Placebo / Oxycodone 30mg: Prior to the experimental conditions, participants will receive non-therapeutic doses of gabapentin 0 mg, p.o., with oxycodone 30 mg, p.o. during a qualifying day session. This session serves as a responsive challenge which is intended to confirm that subjects are able to detect the active drug.
- Placebo / Placebo; Placebo / Oxycodone 20mg; Placebo / Oxycodone 40mg; Gabapentin 600mg / Placebo; Gabapentin 1200mg / Placebo; Gabapentin 600mg / Oxycodone 20mg; Gabapentin 1200mg / Oxycodone 20mg; Gabapentin 600mg / Oxycodone 40mg; Gabapentin 1200mg / Oxycodone 40mg: Participants will receive non-therapeutic experimental doses of gabapentin (0, 600 and 1200 mg, p.o.), alone and in combination with oxycodone (0, 20 and 40 mg, p.o.). The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for gabapentin ≈ 2.5 hr; oxycodone ≈ 1.5 hr). Therefore, oxycodone will be administered 1 hr after gabapentin to align peak responses.
Arm/Group | Pre-Intervention / Days Off | Qualification: Placebo / Oxycodone 30mg | Placebo / Placebo | Placebo / Oxycodone 20mg | Placebo / Oxycodone 40mg | Gabapentin 600mg / Placebo | Gabapentin 1200mg / Placebo | Gabapentin 600mg / Oxycodone 20mg | Gabapentin 1200mg / Oxycodone 20mg | Gabapentin 600mg / Oxycodone 40mg | Gabapentin 1200mg / Oxycodone 40mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 5/11 | 0/11 | 1/11 | 0/11 | 1/11 | 0/11 | 0/11 | 0/11 | 1/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Intervention / Days Off (N=11) | Qualification: Placebo / Oxycodone 30mg (N=11) | Placebo / Placebo (N=11) | Placebo / Oxycodone 20mg (N=11) | Placebo / Oxycodone 40mg (N=11) | Gabapentin 600mg / Placebo (N=11) | Gabapentin 1200mg / Placebo (N=11) | Gabapentin 600mg / Oxycodone 20mg (N=11) | Gabapentin 1200mg / Oxycodone 20mg (N=11) | Gabapentin 600mg / Oxycodone 40mg (N=11) | Gabapentin 1200mg / Oxycodone 40mg (N=11)
Stomachache / upset stomach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea / vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Itching Feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tightness/swollen neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04315181/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04315181/SAP_002.pdf
  • Informed Consent Form (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04315181/ICF_000.pdf